CLINICAL TRIAL: NCT06785181
Title: Dynamic Cardio-, Cerebro-vascular and Cortical Interaction in Healthy Adult Subjects
Brief Title: Dynamic Cardio-vascular, Cerebro-vascular and Cortical Interaction in Healthy Adult Subjects
Acronym: IDEALE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Vlasta Bari, Associate Professor in Bioengineeering, IRCCS Policlinico S. Donato
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IDEALE; 394 (Other: IRCCS Policlinico San Donato)
Record Dates: First submitted 2024-11-04; First posted 2025-01-21 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Cardiac Disease
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HEALTHY SUBJECTS (Experimental): An experimental setup will be devised for the simultaneous monitoring and recording of EEG, ECG, AP, and R together with CBF in healthy volunteers. The experimental protocol including physiological data recordings includes three sessions lasting 10 minutes each: a session at resting state in supine position, a session during autonomic challenge obtained via active standing evoking reflex sympathetic activation, and a session of emotional elicitation via the administration of videos. The overall duration of the experiment is therefore 30 minutes. A total of 40 short video clips of the duration of 15 seconds each will be presented to a total of 50 voluteers will be recruited for the IDEALE study.
  Interventions: Diagnostic Test: Active standing

INTERVENTIONS:
Diagnostic Test: Active standing — a session at resting state in supine position, a session during autonomic challenge obtained via active standing evoking reflex sympathetic activation, and a session of emotional elicitation via the administration of videos
  Other Names: Emotional tests

SUMMARY:
IDEALE aims to assess the status of autonomic function, cerebral autoregulation (CA) and cortical activity in healthy subjects and correlate these functions with the psychological dimension of the subjects.

To this end, parameters of cardiac, cortical, vascular and cerebrovascular variability derived from electrocardiographic, electroencephalographic, respiratory movement, blood pressure, transcranial Doppler signals will be acquired and analysed for each healthy volunteer (TCD) and Laser-Doppler transcutaneous, during a phase of clinostatism (REST) and one of active orthostatism (STAND). In addition, volunteers will be submitted to psychometric tests (Chieti Affective Action Videos, CAAV) to assess the presence of depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* age older than 18 years
* spontaneous sinus rhythm
* signed informed consent

Exclusion Criteria:

* Definite diseases of the Autonomic Nervous System (SNA) or the cardiovascular system
* Central nervous system disorders
* subjects under drug therapy that may affect the cardiovascular system
* pregnancy
* previous diagnosis of depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2027-10-03 (Estimated); Study Completion 2027-10-03 (Estimated)

PRIMARY OUTCOMES:
Autoregulation index (ARI) | 36 months
  ARI is an index describing the state of cerebral autoregulation from mean cerebral blood velocity and mean arterial pressure. Minimum value 0, maximum value 9. ARI>4 means working autoregulation. ARI<4 means impaired autoregulation. It will be computed for all participants.
Baroreflex sensitivity | 36 months
  Baroreflex sensitivity will be measured in ms/mmHg. Minimum value 0. Higher value means a better baroreflex regulation. It will be computed in all participants
Cortical activity | 36 months
  Power of EEG in Alpha and Beta band will be measured in square microvolt. Minimum value 0.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, Milano, Italy

IPD SHARING:
Plan to Share IPD: No